CLINICAL TRIAL: NCT04268472
Title: Bioequivalence Study of GP30101 Film-coated Tablets (LLC "GEROPHARM", Russia) 800 mg Versus Prezista® (Jonson&Jonson, Russia) Film-coated Tablets 800 mg in Healthy Volunteers Under Fed Conditions
Brief Title: Bioequivalence Study of GP30101 800 mg (GEROPHARM) Versus PREZISTA® 800 mg ("Jonson&Jonson", Russia)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GP30101-P4-11
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2020-02

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Darunavir

STUDY DESIGN:
Intervention Model Description: Crossover Assignment two-way crossover
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR Sequence (Experimental): In first Intervention period subjects was administered test medecine (GP30101) and in seconde Intervention period subjects was administered reference medecine (Prezista)
  Interventions: Drug: GP30101; Drug: Prezista®
- RT Sequence (Experimental): In first Intervention period subjects was administered reference medecine (Prezista) and in seconde Intervention period subjects was administered test medecine (GP30101)
  Interventions: Drug: Prezista®; Drug: GP30101

INTERVENTIONS:
Drug: GP30101 — Single oral dose 800 mg, administered in a fed condition, co-administered with low dose ritonavir as a pharmacokinetic enhancer
  Other Names: First aIntervention Period
  Arms: TR Sequence
Drug: Prezista® — Single oral dose 800 mg, administered in a fed condition, co-administered with low dose ritonavir as a pharmacokinetic enhancer
  Other Names: First Intervention Period
  Arms: RT Sequence
Drug: GP30101 — Single oral dose 800 mg, administered in a fed condition, co-administered with low dose ritonavir as a pharmacokinetic enhancer
  Other Names: Second Intervention Period
  Arms: RT Sequence
Drug: Prezista® — Single oral dose 800 mg, administered in a fed condition, co-administered with low dose ritonavir as a pharmacokinetic enhancer
  Other Names: Second Intervention Period
  Arms: TR Sequence

SUMMARY:
Bioequivalence Study of GP30101 800 mg (GEROPHARM) Versus PREZISTA® 800 mg ("Jonson&Jonson", Russia)

DETAILED DESCRIPTION:
Study to evaluate the pharmacokinetic parameters, relative bioavailability and bioequivalence of drugs containing darunavir - GP30101 and Prezista® in healthy volunteers after single orally administered dose, under fed conditions A comparative analysis of adverse events aditionally conducted in this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Male aged 18 to 45 years.
* Verified diagnosis is "healthy" according to data Standard clinical, laboratory and Instrumental methods of examination.
* Body mass index between 18,5 and 30 kg/m2, with body weight 60-100 kg
* Consent to comply with an adequate method of effective contraception throughout the study.
* The consent of volunteers to all restrictions imposed during the study.
* Russian Federation Citizens

Exclusion Criteria:

* History of allergic problems/events.
* Hypersensitivity to heparin, darunavir or any of the excipients of the drugs studied.
* Any acute and chronic diseases, including but not limited to cardiovascular system diseases, bronchopulmonary diseases, neuroendocrine systems diseases, as well as diseases of the gastrointestinal tract, liver, kidneys, blood.
* Positive testing for hepatitis C (antibodies) or hepatitis B (surface antigen), HIV (antibodies to HIV-1/2), syphilis (antibodies to Treponema pallidum).
* The WHO norms deviations of the heart rate (60-89), Sistolic BP (100-130 mm Hg), Diatolic BP (60-89 mm Hg), respiratory rate (12-20), body temperature (35.7 - 37.6 °C).
* Abnormal ECG during screening.
* Inaccessible veins of the upper extremities, vein thrombosis, thrombophlebitis in the anamnesis or in the family history of the next of kin, "compromised" veins due to frequent previous venipuncture.
* Psychiatric disorders, history of epilepsy and seizures.
* Surgical interventions on the gastrointestinal tract (except appendectomy).
* Acute infectious diseases in less than 4 weeks before the start of the study.
* Regular medication use (intake) less than 2 weeks before the start of the study.
* Significant loss of blood within 3 months prior to screening, including but not limited to blood donation or extended surgery or trauma resulting in the blood loss.
* History of alcohol or drugs abuse or any indication of the regular use of more than 10 units of alcohol per week (1 Unit = 200 mL of wine or 500 mL of beer or 50 mL of alcohol 40%).
* Positive test results for alcohol or drug use.
* Nicotine addiction, regular use of tobacco, including all types of electronic cigarettes, less than 6 months prior to screening.
* Participation in a clinical trial of any drugs (including experimental) or experimental medical devices for 3 months or 5 half-lives, whichever is longer, before the study.
* Dehydration due to diarrhea, vomiting, or other causes within the last 24 hours before the start of the study.
* Any diet (for example, vegetarian, fasting, etc.) or lifestyle (including night work and extreme physical activity) that may interfere with the study.
* Taking medications that have a pronounced effect on hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) less than 30 days before the start of the study.
* Volunteers who are obvious or likely, according to the investigator, are unable to understand and evaluate the information on this study as part of the process of signing informed consent, in particular regarding the expected risks and possible discomfort.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
C(max) | -35 min prior dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour post-dose
  Pharmacokinetics by Assessment of Observed Maximum Plasma Concentration (Cmax)
AUC(0-t) | -35 min prior dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour post-dose
  Pharmacokinetics by Assessment of Area Under the Curve From Time Zero Extrapolated to "t" (AUC(0-t)

SECONDARY OUTCOMES:
T(max) | -35 min prior dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour post-dose
  Pharmacokinetics by Assessment of Time of Maximum concentration observed (T(max)
T(1/2) | -35 min prior dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour post-dose
  Pharmacokinetics by Assessment of elimination half-life T(1/2)
K(e) | -35 min prior dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour post-dose
  Pharmacokinetics by Assessment of elimination rate constant

CONTACTS AND LOCATIONS:
Locations (1):
- Yarosslavl Clinical Hospital #3, Yaroslavl, Russia

IPD SHARING:
Plan to Share IPD: No